# Project Title: Testing Self-Control as a Behavior Change Mechanism to Increase Physical Activity

NCT04522141

Informed Consent Upload Date: 03/11/2022 Document Date: 03/17/2020



# Informed Consent Script – Self-Control Intervention Group

You are invited to participate in a research study being conducted by Dr. Mirjam Stieger, a Postdoctoral Associate at Brandeis University. The study is being conducted under the supervision of Dr. Margie E. Lachman, Professor of Psychology.

Please listen to this consent form carefully before you decide whether you want to participate in this research study. We encourage you to ask questions if you want more information about any part of the form or the study.

If you decide to participate in this study you will be asked to sign this form. A copy of the form was sent to you to keep for your records – it has important information, including whom to contact if you have questions in the future.

# What is this study about?

The goal of this study is to investigate daily physical activity in working adults.

## What will you be asked to do if you participate?

We developed the smartphone application MINDHIKE. MINDHIKE will be your personal companion app throughout the study. The study includes three components:

- **Fitbit Step Counter:** You will receive a Fitbit step counter and will be asked to wear it during 12 weeks. You can keep the Fitbit after study completion.
- MINDHIKE Smartphone Application (for free): You will receive a self-control intervention that will help you to increase your physical activity via the MINDHIKE application. The app will remind you to wear the Fitbit step counter each morning and will prompt you for another short (2-3 minutes) coaching session each day.
- Online Questionnaires: You will be asked to answer online questionnaires each Sunday. You will receive the weblink to these questionnaires via the MINDHIKE application.

In total, the study will last over 12 weeks. See below for the detailed study procedure. All study components can be completed flexibly from home so you do not have to come to Brandeis University.

## What is the procedure of the study?

First, you will be asked to fill in a short **screening questionnaire** so we can make sure you meet all our study criteria.

After that, the research team will ship a Fitbit, instruction material. A research assistant will call you to receive informed consent and to personally help you with **installing the smartphone application** MINDHIKE on your own smartphone. You will need to use the MINDHIKE application during the study. The application will remind you every morning to wear your Fitbit and you will have an additional short interaction with the application each day (only 2-3 minutes). You can do this at times that are convenient for you.

At the beginning of the study, you will fill out an **online questionnaire.** This will take you around 30 minutes. You will receive a weblink to this online questionnaire via the MINDHIKE application.

**Week 1:** This week will help you to get used to wearing the Fitbit each day. You will receive a reminder to wear the Fitbit in the morning.

**Weeks 2-8:** During these weeks, you will be asked to wear your Fitbit each day. In addition, you will have another short daily coaching session with the MINDHIKE application (2-3 min). Also, we will ask you to fill in online questionnaires each Sunday. This will take you around 30 minutes. You will receive a weblink to the online questionnaires via the MINDHIKE application.

**Weeks 9-12:** During these weeks, we will ask you to continue wearing your Fitbit. However, you will not have to use the MINDHIKE smartphone application anymore. After these four weeks of waiting period, you will be asked to fill out a last online questionnaire. Please note that for this online questionnaire, we will contact you via E-Mail.



#### What is the benefit of this study?

The self-control intervention may help you to increase your physical activity in daily life and to better understand your daily thoughts, feelings, and behaviors. Moreover, we hope the findings of the study will provide a better understanding of physical activity in working adults.

#### Are there any possible risks to you?

Any risks involved in this study are minimal and no greater than those encountered in everyday life.

#### Will you be compensated or receive anything for participating in the study?

As reimbursement, you can keep the Fitbit after the end of the study. If you stop participating or prefer money, you receive \$1 for each of the 56 first study days and \$14 for participation at the follow-up assessment, totaling to a possible \$70. In addition, as an added incentive, all participants will receive \$25 for completing all aspects of the study.

#### Will it cost you anything to participate in the study?

The only cost to you will be your time. The use of the MINDHIKE application is for free.

## How will your information be kept private?

The information collected by the researchers will be entirely confidential and will be used for research purposes only. Your name will not be used in any reports and collected data will be identified by a number and not your name. Data for all participants will be combined and analyzed as a group. Therefore, we will not be able to give you specific feedback about your individual results. Upon request, we will be happy to send you a summary of the overall research findings when they are available.

#### What will happen with your information once this research study is complete?

Your information will be de-identified (information that can identify you will be destroyed) and kept indefinitely. Note that, despite our best efforts to hide who you are, someone may still be able to identify you. We may also like to share what we learn with other researchers and, if you agree, to put the de-identified data from the questionnaire into a digital data repository (a place that helps researchers to share on-line with other researchers the information that they learn from their research). This allows other researchers access to the data for use in their own research.

#### What if you don't want to participate or change your mind partway through?

Your participation in this study is voluntary; and you are completely free to withdraw from the study at any time or to refuse to answer any questions, or to decline participation in any component of the study. If you stop participating, you receive \$1 for each of the 56 study days and \$14 for participation at the follow-up assessment, totaling to a possible \$70 as a reimbursement for your participation.

#### Who can you call if you have more questions?

If you have any questions about the research being conducted or your participation in the study, feel free to contact the researchers at 781-736-5005 or stieger@brandeis.edu.

If you have any questions about your rights as a subject in this study, would like to speak with someone other than the researchers about concerns you have about the study, or in the event the researchers cannot be reached, please contact the Brandeis University Human Research Protection Program at 781-736-8133 or irb@brandeis.edu.

# **Subject Consent**

Did you listen carefully to this consent form?

Do you have any questions about the study or the informed consent?

Do you understand that your participation is voluntary and that you may withdraw your participation at any time without penalty?

Do you voluntarily agree to participate in this study?

Do you give your permission to share your de-identified data in a data repository?



#### Informed Consent Script - Control Group

You are invited to participate in a research study being conducted by Dr. Mirjam Stieger, a Postdoctoral Associate at Brandeis University. The study is being conducted under the supervision of Dr. Margie E. Lachman, Professor of Psychology.

Please listen to this consent form carefully before you decide whether you want to participate in this research study. We encourage you to ask questions if you want more information about any part of the form or the study.

If you decide to participate in this study you will be asked to sign this form. A copy of the form was sent to you to keep for your records – it has important information, including whom to contact if you have questions in the future.

#### What is this study about?

The goal of this study is to investigate daily physical activity in working adults.

## What will you be asked to do if you participate?

We developed the smartphone application MINDHIKE. MINDHIKE will be your personal companion app throughout the study. The study includes three components:

- **Fitbit Step Counter:** You will receive a Fitbit step counter and will be asked to wear it during 12 weeks. You can keep the Fitbit after study completion.
- MINDHIKE Smartphone Application (for free): The app will remind you to wear the
  Fitbit step counter each morning and will prompt you for another short (2-3 minutes)
  interaction each day
- Online Questionnaires: You will be asked to answer online questionnaires each Sunday. You will receive the weblink to these questionnaires via the MINDHIKE application.

In total, the study will last over 12 weeks. See below for the detailed study procedure. All study components can be completed flexibly from home so you do not have to come to Brandeis University.

## What is the procedure of the study?

First, you will be asked to fill in a short **screening questionnaire** so we can make sure you meet all our study criteria.

After that, the research team will ship a Fitbit, and instruction material. A research assistant will call you personally to receive your informed consent via phone. Also, the research assistant will help you with **installing the smartphone application** MINDHIKE on your own smartphone. You will need to use the MINDHIKE application during the study. The application will remind you every morning to wear you Fitbit and you will have an additional short interaction with the application each day (only 2-3 minutes). You can do this at times that are convenient for you.

At the beginning of the study, you will fill out an **online questionnaire.** This will take you around 30 minutes. You will receive a weblink to this online questionnaire via the MINDHIKE application.

**Week 1:** This week will help you to get used to wearing the Fitbit each day. You will receive a reminder to wear the Fitbit in the morning.

**Weeks 2-8:** During these weeks, you will be asked to wear your Fitbit each day. In addition, you will have another short daily interaction with the MINDHIKE application (2-3 min). Also, we will ask you to fill in online questionnaires each Sunday. This will take you around 30 minutes. You will receive a weblink to the online questionnaires via the MINDHIKE application.

**Weeks 9-12:** During these weeks, we will ask you to continue wearing your Fitbit. However, you will not have to use the MINDHIKE smartphone application anymore. After these four weeks of waiting period, you will be asked to fill out a last online questionnaire. Please note that for this online questionnaire, we will contact you via E-Mail.



## What is the benefit of this study?

You may benefit from tracking your daily activity with the Fitbit. Also, we hope the findings of the study will provide a better understanding of physical activity in working adults.

# Are there any possible risks to you?

Any risks involved in this study are minimal and no greater than those encountered in everyday life.

Will you be compensated or receive anything for participating in the study?

As reimbursement, you can keep the Fitbit after the end of the study. If you stop participating or prefer money, you receive \$1 for each of the 56 first study days and \$14 for participation at the follow-up assessment, totaling to a possible \$70. In addition, as an added incentive, all participants will receive \$25 for completing all aspects of the study.

#### Will it cost you anything to participate in the study?

The only cost to you will be your time. The use of the MINDHIKE application is for free.

#### How will your information be kept private?

The information collected by the researchers will be entirely confidential and will be used for research purposes only. Your name will not be used in any reports and collected data will be identified by a number and not your name. Data for all participants will be combined and analyzed as a group. Therefore, we will not be able to give you specific feedback about your individual results. Upon request, we will be happy to send you a summary of the overall research findings when they are available.

#### What will happen with your information once this research study is complete?

Your information will be de-identified (information that can identify you will be destroyed) and kept indefinitely. Note that, despite our best efforts to hide who you are, someone may still be able to identify you. We may also like to share what we learn with other researchers and, if you agree, to put the de-identified data from the questionnaire into a digital data repository (a place that helps researchers to share on-line with other researchers the information that they learn from their research). This allows other researchers access to the data for use in their own research.

#### What if you don't want to participate or change your mind partway through?

Your participation in this study is voluntary; and you are completely free to withdraw from the study at any time or to refuse to answer any questions, or to decline participation in any component of the study. If you stop participating, you receive \$1 for each of the 56 study days and \$14 for participation at the follow-up assessment, totaling to a possible \$70 as a reimbursement for your participation.

#### Who can you call if you have more questions?

If you have any questions about the research being conducted or your participation in the study, feel free to contact the researchers at 781-736-5005 or stieger@brandeis.edu.

If you have any questions about your rights as a subject in this study, would like to speak with someone other than the researchers about concerns you have about the study, or in the event the researchers cannot be reached, please contact the Brandeis University Human Research Protection Program at 781-736-8133 or irb@brandeis.edu.

#### **Subject Consent**

Did you listen carefully to this consent form?

Do you have any questions about the study or the informed consent?

Do you understand that your participation is voluntary and that you may withdraw your participation at any time without penalty?

Do you voluntarily agree to participate in this study?

Do you give your permission to share your de-identified data in a data repository?